CLINICAL TRIAL: NCT02946853
Title: Junctional AV Ablation in CRT-D Patients With Atrial Fibrillation (JAVA-CRT Trial)
Brief Title: Junctional AV Ablation in CRT-D: JAVA-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jonathan Steinberg, Professor of Medicine - Cardiology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSRB00060626
Record Dates: First submitted 2016-10-24; First posted 2016-10-27 (Estimated); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Systolic Heart Failure; Atrial Fibrillation (Permanent)
Keywords: Atrial Fibrillation; CRT; AV Junction Ablation; LVESV
MeSH Terms: conditions — Heart Failure, Systolic; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRT-D (Active Comparator): Patients will be randomized at enrollment. Patients in this arm of the study will receive cardiac resynchronization therapy with defibrillator (CRT-D).
  Interventions: Device: Cardiac resynchronization therapy - defibrillator
- CRT-D and AVJ Ablation (Experimental): Patients in this arm of the study will receive CRT-D and undergo atrioventricular junctional (AVJ) ablation.
  Interventions: Procedure: Atrioventricular junctional (AVJ) ablation; Device: Cardiac resynchronization therapy - defibrillator

INTERVENTIONS:
Procedure: Atrioventricular junctional (AVJ) ablation — RF energy delivery to AV node to create complete AV block
  Arms: CRT-D and AVJ Ablation
Device: Cardiac resynchronization therapy - defibrillator — Insertion of device capable of providing biventricular pacing and cardiac defibrillation
  Other Names: CRT-D

SUMMARY:
Cardiac resynchronization therapy (CRT) is a demonstrably effective device intervention for patients with heart failure with reduced ejection fraction and specific indication. However, many patients with heart failure (HF) are unable to maintain sinus rhythm and approximately 30-36% of CRT patients are in atrial fibrillation (AF).

DETAILED DESCRIPTION:
This study is designed to evaluate if patients with AF indicated for CRT will have significant reduction in left ventricular end-systolic volume when randomized to atrioventricular junction (AVJ) ablation. In this study, subjects will be randomized to receive CRT-D or CRT-D with AVJ ablation. Randomization will be stratified by enrolling center (1:1 ratio).

ELIGIBILITY:
Inclusion Criteria:

* Optimal pharmacologic therapy is defined by published guidelines from the American Heart Association and the American College of Cardiology
* Initial implantation of CRT-D or prior implantation of CRT-D within one year
* Ischemic or nonischemic cardiomyopathy
* LVEF ≤ 35%
* NYHA class II-IV (ambulatory)
* QRS ≥ 120 ms for LBBB and ≥ 150 ms for non-LBBB patients
* Continuous AF > 3 months when no further efforts to restore sinus rhythm are feasible or pursued

Exclusion Criteria:

* Ventricular rate > 110 bpm at rest despite maximal medical therapy
* Ventricular rate < 50 bpm at rest
* Heart block/symptomatic bradycardia that necessitates permanent pacing
* Acute coronary syndrome or coronary artery bypass surgery within 12 weeks
* Severe aortic or mitral valvular heart disease
* Prior AVJ ablation
* Any medical condition likely to limit survival to < 1 year
* Patients with ACC/AHA Stage D refractory Class IV symptoms listed for transplant or requiring inotropic support
* Contraindication to systematic anticoagulation
* Renal failure requiring dialysis
* AF due to reversible cause e.g. hyperthyroid state
* Pregnancy
* Participation in other clinical trials that will affect the objectives of this study
* History of non-compliance to medical therapy
* Inability or unwillingness to provide informed consent
* Patients with short-lived AF or those in sinus rhythm are ineligible

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Steinberg, MD, Principal Investigator — University of Rochester
Locations (21):
- United States (21):
  - Arkansas Cardiology, Little Rock, Arkansas
  - Huntington Memorial Hospital, Pasadena, California
  - Emory Healthcare, Atlanta, Georgia
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - University of Iowa, Iowa City, Iowa
  - Lahey Clinic, Burlington, Massachusetts
  - University of Massachusetts-Worchester, Worcester, Massachusetts
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Catholic Medical Ctr/New England Heart-Vasc Inst, Manchester, New Hampshire
  - SUNY at Buffalo, Buffalo, New York
  - Northwell Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Oregon Health & Science University, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - INOVA, Woodbridge, Virginia
  - Kootenai Heart Clinics, LLC, Spokane, Washington
  - Multicare Institute for Research and Innovation, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steinberg JS, Gorcsan J, Mazur A, Jain SK, Rashtian M, Greer GS, Zarraga I, Vloka M, Cook MM, Salam T, Mountantonakis S, Beck H, Silver J, Aktas M, Henrikson C, Schaller RD, Epstein AE, McNitt S, Schleede S, Peterson D, Goldenberg I, Zareba W. Junctional AV ablation in patients with atrial fibrillation undergoing cardiac resynchronization therapy (JAVA-CRT): results of a multicenter randomized clinical trial pilot program. J Interv Card Electrophysiol. 2022 Aug;64(2):519-530. doi: 10.1007/s10840-021-01116-6. Epub 2022 Jan 18. PMID 35043250

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CRT-D | CRT-D and AVJ Ablation
Started | 13 | 13
Completed | 12 | 13
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRT-D | CRT-D and AVJ Ablation | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Full Range); unit: years] | 72 [66 to 78] | 73 [65 to 81] | 73 [65 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 10 | 9 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11 | 13 | 24
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
LV End Systolic Volume [Mean (Standard Deviation); unit: cc] | 115 (29) | 121 (39) | 118 (30)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Reduction ≥ 15% in Left Ventricular End-systolic Volume (LVESV)
Description: Number of patients with reduction ≥ 15% in left ventricular end-systolic volume (LVESV) in each arm of the study.
Time Frame: Baseline to 6 months
Population: Some patients did not undergo outcome measures due to inability to come for follow-up due to COVID-19.
Measure: Count of Participants; unit: Participants
Arm/Group | CRT-D | CRT-D and AVJ Ablation
Number analyzed (Participants) | 10 | 12
Participants | 5 | 6
Statistical Analysis 1: Comparison: CRT-D vs CRT-D and AVJ Ablation; Test type: Superiority; p = 1.00, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.14 to 7.21]

2. Secondary Outcome: Change in Left Ventricular Ejection Fraction (EF)
Description: Change in left ventricular ejection fraction from baseline to 6 months. Units are expressed in percent and change may vary from -20% to 20%. More negative numbers are desired representing improvement from baseline to 6 months.
Time Frame: Baseline to 6 months
Population: A small number patients were unable to return for follow-up due the the outbreak of COVID-19 and some outcome measures were not completed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | CRT-D | CRT-D and AVJ Ablation
Number analyzed (Participants) | 10 | 12
percentage | -7.0 (11.8) | -8.6 (9.1)
Statistical Analysis 1: Comparison: CRT-D vs CRT-D and AVJ Ablation; Test type: Superiority; p = 0.974, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -1.0

3. Other Pre Specified Outcome: Percent Change in Left Ventricular End-diastolic Volume (LVEDV)
Description: Percent change in left ventricular end-diastolic volume (LVEDV) by study arm.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: % change in volume
Arm/Group | CRT-D | CRT-D and AVJ Ablation
Number analyzed (Participants) | 12 | 10
% change in volume | -1.1 (23.7) | -3.5 (13.2)
Statistical Analysis 1: Comparison: CRT-D vs CRT-D and AVJ Ablation; Some patients did not undergo 6 month echocardiogram due to restrictions related to COVID-19; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.5

4. Other Pre Specified Outcome: Number of Patients With Heart Failure Hospitalizations
Description: Number of patients with heart failure hospitalizations in each arm of the study.
Time Frame: Baseline to 6 months
Measure: Number; unit: participants
Arm/Group | CRT-D | CRT-D and AVJ Ablation
Number analyzed (Participants) | 13 | 13
participants | 1 | 1
Statistical Analysis 1: Comparison: CRT-D vs CRT-D and AVJ Ablation; Test type: Superiority; p = 1.00, Fisher Exact; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.1 to 84.4]

5. Other Pre Specified Outcome: Number of Patients With Implantable Cardioverter-defibrillator Delivered Inappropriate Therapy
Description: Number of patients with implantable cardioverter-defibrillator delivered inappropriate therapy in each arm of the study
Time Frame: Baseline to 6 months
Measure: Number; unit: participants
Arm/Group | CRT-D | CRT-D and AVJ Ablation
Number analyzed (Participants) | 13 | 13
participants | 0 | 0
Statistical Analysis 1: Comparison: CRT-D vs CRT-D and AVJ Ablation; Test type: Superiority; p = 1.00, Fisher Exact; Odds Ratio (OR) = 1.00

6. Other Pre Specified Outcome: Number of Patients With Implantable Cardioverter-defibrillator Delivered Appropriate Therapy for VT or VF
Description: Number of patients with implantable cardioverter-defibrillator delivered appropriate therapy treatment by ICD for VT/VF in each arm of the study.
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CRT-D | CRT-D and AVJ Ablation
Number analyzed (Participants) | 13 | 13
Participants | 1 | 0
Statistical Analysis 1: Comparison: CRT-D vs CRT-D and AVJ Ablation; Test type: Superiority; p = 1.00, Fisher Exact; Odds Ratio (OR) = 0, 95% CI 2-sided [0.00 to 42.00]

7. Other Pre Specified Outcome: Percentage of Biventricular Pacing
Description: Amount of time that CRT is delivered
Time Frame: At 6 months
Measure: Mean (Standard Deviation); unit: % BiV pacing
Arm/Group | CRT-D | CRT-D and AVJ Ablation
Number analyzed (Participants) | 13 | 13
% BiV pacing | 77.1 (26.3) | 97.7 (3.6)
Statistical Analysis 1: Comparison: CRT-D vs CRT-D and AVJ Ablation; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 20.6

8. Other Pre Specified Outcome: Kansas City Cardiomyopathy Questionnaire
Description: Scoring scale from 0 to 100. Higher scores represent better quality of life.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CRT-D | CRT-D and AVJ Ablation
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline | 56.6 (17.6) | 61.9 (26.9)
  6 months | 69.1 (20.3) | 81.3 (18.2)
Statistical Analysis 1: Comparison: CRT-D vs CRT-D and AVJ Ablation; Test type: Superiority; p = 0.565, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 23.7

9. Other Pre Specified Outcome: Number of Participants With Episodes of Ventricular Fibrillation Following AV Junctional Ablation as Detected on ICD
Description: Episodes of ventricular fibrillation following AV junctional ablation as detected on ICD in each arm of the study.
Time Frame: Baseline to one month
Measure: Number; unit: participants
Arm/Group | CRT-D | CRT-D and AVJ Ablation
Number analyzed (Participants) | 13 | 13
participants | 1 | 0
Statistical Analysis 1: Comparison: CRT-D vs CRT-D and AVJ Ablation; Test type: Superiority; p = 1.00, Fisher Exact; Odds Ratio (OR) = 0, 95% CI 2-sided [0.0 to 42.0]

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Arm/Group | CRT-D | CRT-D and AVJ Ablation
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT-D (N=13) | CRT-D and AVJ Ablation (N=13)
Hospitalization with heart failure (Cardiac disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The study results were hampered by difficulty meeting the sample size targets, resulting in lower than planned power and precision. In addition, the trial did not have a study arm without any intervention (either CRT or AVJA) so that "untreated" patients could be compared to each intervention group. Hard clinical endpoints including hospitalization, death and ICD events were too infrequent to make meaningful comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT02946853/Prot_SAP_000.pdf